BeiGene 09 February 2023

NCT03666143



# STATISTICAL ANALYSIS PLAN

**Study Protocol Number:** BGB-900-103

Study Protocol Title: A Phase 1b Study to Assess the Safety, Tolerability,

Pharmacokinetics, and Preliminary Antitumor Activity of Sitravatinib in Combination with Tislelizumab in Patients with

**Advanced Solid Tumors** 

**Date:** 09 February 2023

Version: 1.0

BeiGene 09 February 2023

# SIGNATURE PAGE

| Author: | |
|---------|-----------------------------------------|
| | Signature |
| | Date: <u>09-Feb-2023 </u> 05:49:22 PST |

# Approval



| BGB-900-103 |
|-------------------------------|
| Statistical Analysis Plan 1.0 |

# BeiGene 09 February 2023

| TABLE OF CONTENTS | |
|------------------------------------------------------------------------|-----|
| LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS | 6 |
| 1INTRODUCTION | 8 |
| 2STUDY OVERVIEW | 8 |
| 2.1Study Design | 8 |
| 2.2. Study Assessments. | 10 |
| 3 STUDY OBJECTIVES | 11 |
| 3.1Primary Objective | 11 |
| 3.2Secondary Objective | 11 |
| 3.3. Exploratory Objective | 11 |
| 4 STUDY ENDPOINTS. | 12 |
| 4.1Primary Endpoint(s) | 12 |
| 4.2. Secondary Endpoints | 12 |
| 4.3. Exploratory Endpoints | 12 |
| 5 SAMPLE SIZE CONSIDERATIONS | 13 |
| 6STATISTICAL METHODS | 13 |
| 6.1 Analysis Sets | 13 |
| 6.2Multiplicity Adjustment | 13 |
| 6.3 Data Analysis General Considerations | 14 |
| 6.3.1 Definitions and Computations | 14 |
| 6.3.2Conventions | 14 |
| 6.3.3 Handling of Missing Data | 15 |
| 6.4. Patient Characteristics | 15 |
| 6.4.1 Patient Disposition | 15 |
| 6.4.2 Protocol Deviations | 15 |
| 6.4.3 Demographic and Other Baseline Characteristics | 15 |
| 6.4.4 Disease History | 16 |
| 6.4.5 Prior Anticancer Drug Therapies and Surgeries | 17 |
| 6.4.5.1 Prior Anticancer Drug Therapies | 18 |
| 6.4.5.2 Prior Anticancer Surgeries/ Procedures with Therapeutic Intent | 18 |
| 6.4.5.3 Prior Radiotherapies | 18 |
| 6.4.6 Prior and Concomitant Medications | 1.9 |

| BGB-900-103<br>Statistical Analysis Plan 1.0 | BeiGene 09 February 2023 |
|---|---|
| 6.4.7 Medical History | |
| 6.5 Efficacy Analysis | 18 |
| 6.5.1 Secondary Efficacy Endpoints | 18 |
| 6.5.2 Exploratory Efficacy Endpoints | 21 |
| 6.6. Safety Analysis | 22 |
| 6.6.1 Extent of Exposure | 23 |
| 6.6.2 Adverse Events | 23 |
| 6.6.2.1 Treatment Emergent Adverse Event | 24 |
| 6.6.2.2 Immune- Mediated Adverse Event | 25 |
| 6.6.2.3 Infusion-related Adverse Event | 26 |
| 6.6.2.4 Death | 26 |
| 6.6.3 Laboratory Values | 26 |
| 6.6.4 Vital Signs | 28 |
| 6.6.5 Electrocardiograms (ECG) | 28 |
| 6.6.6 Eastern Cooperative Oncology Group (ECOG) Performance Status | 28 |
| 6.7 Pharmacokinetic Analysis | 28 |
| 6.7.1 Pharmacokinetic Analysis of Sitravatinib | 28 |
| 6.7.2 Pharmacokinetic Analysis of Tislelizumab | 29 |
| 6.8Immunogenicity Analysis | 30 |
| 7INTERIM ANALYSIS | 30 |
| 8 CHANGES IN THE PLANNED ANALYSIS | 30 |
| 9REFERENCES | 32 |
| APPENDIX 1. IMPUTATION OF MISSING OR PARTIALLY MISSING DA | ATES33 |
| 1.1 Prior/Concomitant Medications/Procedures | 33 |
| 1.2 Adverse Events | 33 |
| 1.3 Disease history and prior therapy (Drug, surgery/procedure, radiotherapy) | |
| 1.4 Subsequent anti-cancer therapy | 35 |
| APPENDIX 2 PLUES FOR IDENTIFYING MISSING TUMOR ASSESSME | INTS 36 |

BeiGene 09 February 2023

# LIST OF TABLES

| Table 1: Censoring Rules for Progression-Free Survival Per RECIST Version 1.1 | 19 |
|---|---|
| Table 2: Measurement of CA-125 | 22 |
| Table 3: Clinical Laboratory Assessment | 27 |
| Table 4: Statistical Analysis Plan Changes | 31 |
| Table 5: Example of Scheduled Tumor Assessments With Time Window | 36 |

BeiGene 09 February 2023

# LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

| Abbreviation | Definition |
|---|---|
| ADA | Antidrug Antibody |
| AE | Adverse Event |
| ATC | Anatomical Therapeutic Chemical |
| BLQ | Below the Assay Quantification Limit |
| C1D1 | Cycle 1 Day 1 |
| C1D21 | Cycle 1 Day 21 |
| CA-125 | Cancer Antigen 125 |
| CBR | Clinical Benefit Rate |
| CI | Confidence Interval |
| CR | Complete Response |
| CV | Coefficient of Variance |
| DCR | Disease Control Rate |
| DOR | Duration of Response |
| ECG | Electrocardiograms |
| ECOG | Eastern Cooperative Oncology Group |
| GCIG | Gynecologic Cancer Intergroup |
| imAE | Immune-mediated AE |
| IRR | Infusion-related Reaction |
| MedDRA | Medical Dictionary for Regulatory Activities |
| NA | Not Assessable |
| NCI-CTCAE | National Cancer Institute Common Terminology Criteria for Adverse Events |
| NSCLC | Non-Small Cell Lung Cancer |
| OC | Ovarian Cancer |
| ORR | Objective Response Rate |
| OS | Overall Survival |
| PD | Progressive Disease |
| PD-1 | Programmed Cell Death Protein-1 |
| PD-L1 | Programmed Cell Death Protein-Ligand 1 |
| PFS | Progression-Free Survival |
| PGx | Pharmacogenetic |
| PK | Pharmacokinetic(s) |
| PR | Partial Response |
| PT | Preferred Term |
| RCC | Renal Cell Carcinoma |
| RECIST | Response Evaluation Criteria in Solid Tumors |
| SAE | Serious Adverse Event |

BeiGene 09 February 2023

| SD | Stable Disease |
|--------|-------------------------------------------|
| SFD | Study Follow-up Duration |
| SOC | System Organ Class |
| TEAE | Treatment-Emergent Adverse Event |
| TTR | Time to Response |
| WHO DD | World Health Organization Drug Dictionary |

BeiGene 09 February 2023

#### 1. INTRODUCTION

The purpose of this statistical analysis plan (SAP) is to describe the procedures and the statistical methods that will be used to analyze and report results for BGB-900-103: a Phase 1b study to assess the safety, tolerability, pharmacokinetics, and preliminary antitumor activity of sitravatinib in combination with tislelizumab in patients with advanced solid tumors. The focus of this SAP is for the planned final analysis specified in the study protocol. The analysis details for Pharmacodynamics, Pharmacogenomics and Biomarker are not described within this SAP. Separate analysis plans will be completed for these analyses and will be attached in addition to this SAP to the clinical study report.

## 2. STUDY OVERVIEW

# 2.1. Study Design

This is an open-label, multicenter, non-randomized Phase 1b clinical study for patients with histologically or cytologically confirmed locally advanced or metastatic tumors including non-squamous or squamous non-small cell lung cancer (NSCLC), renal cell carcinoma (RCC), epithelial ovarian cancer (OC), or melanoma.

All patients will receive sitravatinib 120 mg orally, once daily in combination with tislelizumab 200 mg intravenously once every 3 weeks until occurrence of progressive disease (PD), unacceptable toxicity, death, withdrawal of consent, or study termination by sponsor.

There will be a total of 9 cohorts in the study. Approximately 60 patients will be enrolled into Cohort E, including at least 20 patients who failed the prior bevacizumab treatment and at least 20 patients will be Caucasian. In addition, approximately 20 patients will be enrolled into each of the rest of the cohorts. The patients will be enrolled according to their tumor type and prior anti-programmed cell death protein-1 (PD-1)/programmed cell death protein ligand-1 (PD-L1) antibody treatment.

- Cohort A: Anti-PD-1/PD-L1 antibody refractory/resistant metastatic, non-squamous NSCLC
- Cohort B: Anti-PD-1/PD-L1 antibody naïve metastatic, non-squamous NSCLC
- Cohort C: Anti-PD-1/PD-L1 antibody refractory/resistant metastatic or advanced RCC
- Cohort D (China-only): Metastatic or advanced RCC without prior systemic therapy
- Cohort E: Anti-PD-1/PD-L1 antibody naïve recurrent and platinum-resistant epithelial OC
- Cohort F: Anti-PD-1/PD-L1 antibody refractory/resistant metastatic, squamous NSCLC
- Cohort G: Anti-PD-1/PD-L1 antibody refractory/resistant unresectable or metastatic melanoma
- Cohort H: PD-L1 positive, locally advanced or metastatic, non-squamous NSCLC without prior systemic treatment in metastatic setting
- Cohort I: PD-L1 positive, locally advanced or metastatic, squamous NSCLC without prior systemic treatment in metastatic setting

The study schema is in Figure 1.

BeiGene 09 February 2023

Figure 1. Study Schema



Abbreviations: IHC, immunohistochemistry; mNSCLC, metastatic non-small cell lung cancer; mRCC, metastatic renal cell carcinoma; NSCLC, non-small cell lung cancer; OC, ovarian cancer; PD, progressive disease; PD-1, programmed cell death protein-1; PD-L1, programmed cell death protein ligand-1; RCC. renal cell carcinoma; RECIST, Response Evaluation Criteria in Solid Tumors; VEGF, Vascular endothelial growth factor; VEGFR TKI, vascular endothelial growth factor receptor tyrosine kinase inhibitors.

Key changes made from original protocol 0.0 (26 June 2018) to protocol amendment 1.0 (02 March 2019) were as follows.

- Added Cohort F of squamous NSCLC patients.
- Added Cohort G of melanoma patients.

Key changes made from protocol amendment 1.0 (02 March 2019) to protocol amendment 2.0 (12 June 2019) were as follows.

- Added Cohort H for PD-L1 positive, non-squamous locally advanced or metastatic NSCLC without prior systemic treatment in metastatic setting.
- Added Cohort I for PD-L1 positive, locally advanced or metastatic squamous NSCLC without prior systemic treatment in metastatic setting.

Key changes made from protocol amendment 2.0 (12 June 2019) to protocol amendment 3.0 (04 November 2019) were as follows.

- Increase sample size to 60 subjects in Cohort E.
- Revised the subject type of Cohort F.
  - Revise the definition of Cohort F: anti-PD-1/PD-L1 antibody refractory/resistant metastatic, squamous NSCLC.
  - o Add the definition to clarify "anti-PD-1/PD-L1 antibody refractory/resistant metastatic, squamous NSCLC" in Cohort F.

Cohort F will only enroll prior anti-PD-1/PD-L1 antibody refractory/resistant squamous NSCLC until the total number of prior anti-PD-1/PD-L1 antibody treated squamous NSCLC reaches 20 patients. The prior anti-PD-1/PD-L1 naïve patients who enrolled before the amendment can continue their treatment per the protocol. It is to further investigate the safety and efficacy for patients with anti-PD-1/PD-L1 antibody treated squamous NSCLC. The anti-PD-1/PD-L1 antibody naïve patient will be no longer enrolled in this cohort after this amendment is effective.

#### Note

The below definition clarifies "anti-PD-1/PD-L1 antibody refractory/resistant" in Cohort A, C and F.

Radiographic progression per RECIST v1.1 on or after anti-PD-1/PD-L1-containing therapy as the most recent treatment with best response defined as follows.

- a. Resistant (i.e., RECIST v1.1-defined partial response (PR), complete response (CR), or stable disease (SD) for at least 12 weeks after initiation of treatment followed by radiographic progression of disease)
- b. Refractory (i.e., radiographic progression of disease < 12 weeks after initiation of treatment)

The below definition clarifies "anti-PD-1/PD-L1 antibody refractory/resistant" in Cohort G.

Radiographic disease progression per RECIST v1.1 on or after the immediate prior first line anti-PD-1/PD-L1 monotherapy. If adjuvant, disease progression within 6 months of last dose of anti-PD-1 therapy.

- a. Resistant (ie, RECIST v1.1 defined partial, complete response or stable disease for at least 12 weeks after initiation of treatment followed by radiographic progression of disease) If treated with anti-PD-1/PD-L1 adjuvant therapy, patient relapses while on treatment or within 6 months after last dose of anti-PD-1/PD-L1 therapy is also considered resistant.
- b. Refractory (ie, radiographic progression of disease < 12 weeks after initiation of treatment).

# 2.2. Study Assessments

**Tumor Assessment** 

Tumor assessments will be performed by investigator using Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1 criteria (Eisenhauer EA, 2009). For ovarian cancer patients, response will be assessed using RECIST v1.1 and the Gynecologic Cancer Intergroup (GCIG) working group criteria). Tumor imaging will be performed at baseline (within 28 days prior to the first dose of study drugs). During the study, tumor imaging will be performed approximately every 6 weeks ( $\pm$  7 days) in the first 12 months and thereafter approximately every 9 weeks ( $\pm$  7 days). If a patient discontinues study treatment due to any reasons other than disease progression, tumor assessments will continue to be performed as scheduled until initiation of a new anticancer therapy, disease progression, loss to follow up, withdrawal of consent, death, or until the study terminates, whichever occurs first.

## Safety Assessment

Patients will be evaluated for any adverse events (AEs) and serious adverse events (SAEs) occurring up to 30 days after the last dose of study drugs (all severity grades, per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0) or initiation of a new anticancer therapy, whichever occurs first, and immune-mediated AEs (imAEs) occurring up to 90 days after the last dose of tislelizumab regardless of initiation of a subsequent anticancer therapy. At the end of treatment, ongoing AEs considered related to study treatment will be followed until the event has resolved to baseline or  $\leq$  Grade 1, the event is assessed by the investigator as stable, the patient is lost to follow-up, the patient withdraws consent, or it has been determined that study treatment or participation is not the cause of the AE. All drug-related SAEs will be recorded by investigator after treatment discontinuation until patient death, withdrawal of consent, or loss to follow up, whichever occurs first.

## 3. STUDY OBJECTIVES

# 3.1. Primary Objective

• To characterize safety and tolerability of sitravatinib in combination with tislelizumab

# 3.2. Secondary Objective

- To assess the preliminary antitumor activity of sitravatinib in combination with tislelizumab
- To characterize the Pharmacokinetic (PK) profiles of sitravatinib after single dose and at steady state when given in combination with tislelizumab

# 3.3. Exploratory Objective

- To assess PK and immunogenicity of tislelizumab when given in combination with sitravatinib
- To explore potential pharmacodynamic biomarkers for sitravatinib in combination with tislelizumab
- To explore potential biomarkers of efficacy, resistance, or PD in tumor tissue and in peripheral whole blood
- To assess overall survival (OS)

- To explore effect of pharmacogenetic (PGx) polymorphisms on PK of sitravatinib
- To assess the preliminary antitumor activity of sitravatinib in combination with tislelizumab for ovarian cancer patients based on the GCIG working group criteria

BeiGene

09 February 2023

#### 4. STUDY ENDPOINTS

## 4.1. **Primary Endpoint(s)**

 Safety and tolerability – assessed throughout the study by monitoring AEs and SAEs per NCI-CTCAE version 5.0, relevant physical examination, electrocardiograms, and laboratory assessments as needed

# 4.2. Secondary Endpoints

- Objective response rate (ORR) defined as the percentage of patients whose best overall response (BOR) is CR or PR assessed by investigators per RECIST v1.1
- Duration of response (DOR) defined as the time from the first determination of an objective response until the first documentation of PD as assessed by investigator per RECIST v1.1, or death, whichever comes first
- Disease control rate (DCR) defined as the proportion of patients with BOR as CR, PR, or SD assessed by investigator per RECIST v1.1
- Progression-free survival (PFS) defined as the time from the date of first dose to the date
  of first documentation of PD assessed by the investigator per RECIST v1.1 or death,
  whichever occurs first
- Plasma concentrations of sitravatinib
- Derived PK parameters of single dose sitravatinib
- Derived PK parameters of repeated dose sitravatinib

# 4.3. Exploratory Endpoints

- Serum concentrations of tislelizumab and anti-tislelizumab antibodies
- Changes of potential pharmacodynamic biomarkers in response to sitravatinib in combination with tislelizumab, such as, but not limited to, soluble vascular endothelial growth factor receptor 2 (sVEGFR-2), and immune cell subpopulations in peripheral blood
- Potential biomarkers including but not limited to PD-L1 expression, immune-cell profiling, tumor mutation load and gene expression profiling, and the association with disease status and/or the response to sitravatinib in combination with tislelizumab
- Overall survival (OS) defined as the time from the date of first dose until the date of death due to any cause
- The effect of genetic polymorphisms of hepatic metabolizing enzymes and transporters, including but not limited to CYP1A2, 2D6, and 2C8 on the PK of sitravatinib
- Efficacy evaluations for ovarian cancer patients

 ORR per CA-125 – defined as the proportion of patients who have confirmed CR or PR by the investigator's review per cancer-antigen 125 (CA-125) (GCIG working group criteria)

o PFS per CA-125 – defined as the time from the date of first dose to the date of first documentation of PD assessed by the investigator per CA-125 (GCIG working group criteria) or death, whichever occurs first in all patients with ovarian cancer (cohort E)

### 5. SAMPLE SIZE CONSIDERATIONS

Based on the protocol amendment 3.0, approximately 220 to 240 patients (approximately 60 patients for cohort E, and 20 patients for each of the rest of the cohorts) are expected to be enrolled to analyze safety and preliminary efficacy for sitravatinib plus tislelizumab. Of the approximately 60 patients enrolled into cohort E, at least 20 patients who failed the prior bevacizumab treatment and at least 20 patients will be Caucasian. Enrollment into these cohorts will occur simultaneously, independently of each other.

### 6. STATISTICAL METHODS

# 6.1. Analysis Sets

The Safety Analysis Set includes all patients who received any dose of any study drug. The Safety Analysis Set is used for all primary safety and efficacy analysis except for the response analysis.

The Efficacy Evaluable Analysis Set consists of all treated patients in the Safety Analysis Set with measurable baseline assessment per RECIST 1.1 who had at least one evaluable post-baseline tumor assessment unless treatment was discontinued due to clinical disease progression or early death (within 13 weeks of the first dose date). The Efficacy-Evaluable Analysis Set will be used for primary response analysis.

The Evaluable for CA-125 Response Set is defined as the subset of subjects in the safety population in cohort E with baseline CA-125  $\geq$  2 x ULN (GCIG working group criteria). This is the primary analysis set for the analysis of CA-125 response rate in cohort E.

**The Sitravatinib Pharmacokinetic Analysis Set** includes all patients who contributed at least 1 quantifiable PK sample for sitravatinib. The sitravatinib pharmacokinetic analysis set will be used for PK analysis for sitravatinib.

**The Tislelizumab Pharmacokinetic Analysis Set** includes all patients who contributed at least 1 quantifiable PK sample for tislelizumab. The Tislelizumab Pharmacokinetic Analysis Set will be used for PK analysis for tislelizumab.

The Tislelizumab Antidrug Antibody (ADA) Analysis Set includes all patients who received at least 1 dose of tislelizumab and for whom both baseline ADA and at least 1 postbaseline ADA results are available. The ADA analysis set will be used for ADA analysis for tislelizumab.

# **6.2.** Multiplicity Adjustment

Since no formal hypothesis is tested in this study, multiplicity adjustment is not needed.

## 6.3. Data Analysis General Considerations

### **6.3.1.** Definitions and Computations

### Study drugs

Study drugs include tislelizumab and sitravatinib. Tislelizumab (200 mg) will be administered on Day 1 of each 21-day cycle (every 3 weeks). Sitravatinib capsules will be administered orally, once daily continuously for a total daily dose of 120 mg.

#### Study day

Study day will be calculated in reference to the date of the first dose of study drug for both safety analysis and efficacy analysis. For assessments conducted on or after the date of first dose of study drug, the study day will be calculated as (assessment date – date of first dose of study drug + 1). For assessments conducted before the date of first dose of study drug, study day is calculated as (assessment date – date of first dose of study drug). There is no study day 0. In the situation where the event date is partial or missing, the date will appear partial or missing in the listings. Study day and any corresponding durations will be presented based on the imputations specified in Appendix 1.

### Baseline value

Unless otherwise specified, a baseline value is defined as the last non-missing value collected before the first dose of study drug.

## Study Follow-up Duration

Study follow-up duration (SFD) is defined as the time from the first dose date to the death date or study discontinuation date (whichever occurs first) for patients discontinued from the study, or the data cutoff date for patients continuing in the study.

All calculations and analyses will be conducted using SAS® Version 9.4 or higher.

#### 6.3.2. Conventions

No formal hypothesis will be tested in this study. Data will be mainly analyzed descriptively. Confidence intervals (CIs) will be constructed to describe the precision of the point estimates of interest (eg, ORR and DCR). Data will be summarized by cohorts for efficacy analysis. And data will be summarized by cohorts, NSCLC population, and total for safety analysis. In tables and figures, cohort F only includes patients with anti-PD-1/PD-L1 antibody refractory/resistant, metastatic, squamous NSCLC per protocol amendment (PA) 3.0, and NSCLC population and total includes all the patients who met the inclusion criteria per PA 1.0, PA 2.0, and PA 3.0. In listings, cohort F includes all the patients who met the inclusion criteria of cohort F per PA 1.0, PA 2.0, and PA 3.0. Unless otherwise specified, the following conventions will be applied to all analyses.

- 1 year = 365.25 days. Number of years is calculated as (days/365.25) rounded up to 1 decimal place.
- 1 month = 30.4375 days. Number of months is calculated as (days/30.4375) rounded up to 1 decimal place.
- Age will be calculated as the integer part of (date of informed consent date of birth + 1)/365.25.

- Duration of image-based event endpoints (such as PFS) will be based on the actual date the radiograph was obtained rather than the associated visit date.
- For laboratory results collected in numerical range, if lab results  $\geq x$  then set as x; if  $\leq x$ , then x/2.
- For by-visit observed data analysis, percentages will be calculated based on the number of patients with non-missing data as the denominator, unless otherwise specified.
- For continuous endpoints, summary statistics will include n, mean, standard deviation, median, Q1, Q3 and range (minimum and maximum). For PK concentration and parameters, geometric mean, and geometric coefficient of variance (CV%) will also be included in the summary while Q1 and Q3 may not be calculated.
- For discrete endpoints, summary statistics will include frequencies and percentages.

### 6.3.3. Handling of Missing Data

Missing data will not be imputed unless otherwise specified elsewhere in this SAP. Missing dates or partially missing dates will be imputed conservatively for adverse events and prior/concomitant medications/procedures. Specific rules for the handling of missing or partially missing dates for adverse events and prior/concomitant medications/procedures are provided in Appendix 1. Byvisit endpoints will be analyzed using observed data unless otherwise specified. For observed data analysis, missing data will not be imputed, and only the observed records will be included.

#### 6.4. Patient Characteristics

## 6.4.1. Patient Disposition

The number (percentage) of patients who signed informed consent, enrolled in the study, screen failures, screened previously, and reason for screen failure will be summarized in all patients.

The number (percentage) of patients treated, discontinued from the study, discontinued from the treatment (all treatments), reasons for discontinued from the study, reasons for discontinued from the treatment, and the duration of study follow-up will be summarized in the Safety Analysis Set.

The reasons for patients discontinued from tislelizumab or sitravatinib will be summarized separately in Safety Analysis Set.

Patient data listings of patient disposition will be provided.

#### **6.4.2.** Protocol Deviations

Protocol deviation criteria will be established together with its category/term of important and not important. Patients with important protocol deviations will be identified and documented before the database lock. Important protocol deviations will be summarized for all patients in the Safety Analysis Set. They will also be listed by each category. Multiple deviations within the same category are counted once per patient.

#### 6.4.3. Demographic and Other Baseline Characteristics

Demographics and other baseline characteristics will be summarized using descriptive statistics in the Safety Analysis Set, including the following variables:

• Age (continuously and by categories [ $< 65 \text{ or } \ge 65 \text{ years}$ ])

BeiGene 09 February 2023

- Sex
- Race
- Ethnicity
- Geographic Region
- Weight (kg)
- BMI  $(kg/m^2)$
- ECOG performance status
- Smoking status
- Alcohol consumption
- PD-L1 Tumor Cell Score

## 6.4.4. Disease History

The number (percentage) of patients reporting a history of disease and characteristics, as recorded on the eCRF, will be summarized in the Safety Analysis Set.

Disease history of NSCLC includes the following characteristics:

- Disease stage at initial diagnosis
- Patients with metastatic disease at study entry
- Time from initial diagnosis to time of diagnosis of metastatic disease/locally advanced disease
- Time from diagnosis of metastatic disease/locally advanced disease to first dose date
- Known metastatic site at study entry
- Histology/Cytology
- TNM staging at initial diagnosis

Disease history of Epithelial OC includes the following characteristics:

- Disease stage at initial diagnosis
- Patients with metastatic disease at study entry
- Time from initial diagnosis to time of diagnosis of metastatic disease/ locally advanced disease
- Time from diagnosis of metastatic disease/locally advanced disease to first dose date
- Known metastatic site at study entry
- Epithelial type
- Histologic grade
- Primary location

BeiGene 09 February 2023

• TNM staging at initial diagnosis

Disease history of RCC includes the following characteristics:

- Disease stage at study entry
- Disease stage at initial diagnosis
- Patients with metastatic disease at study entry
- Time from initial diagnosis to time of diagnosis of metastatic disease/ locally advanced disease
- Time from diagnosis of metastatic disease/locally advanced disease to first dose date
- Known metastatic site at study entry
- Histology/Cytology
- AJCC grade
- Prognostic risk groups at study entry
- Risk models
- Status of primary tumor at study entry
- TNM staging at initial diagnosis

Disease history of Melanoma includes the following characteristics:

- Disease stage at initial diagnosis
- Patients with metastatic disease at study entry
- Time from initial diagnosis of metastatic disease/locally advanced disease to first dose date
- Time from diagnosis of metastatic disease/locally advanced disease to first dose date
- Known metastatic site at study entry
- Histology/Cytology
- Primary Location
- BRAF Mutation Status
- TNM staging at initial diagnosis

The listings of disease history and characteristic with different indications will be provided.

### 6.4.5. Prior Anticancer Drug Therapies and Surgeries

Prior anticancer drug therapies, prior anticancer surgeries/ procedures with therapeutic intent, and prior radiotherapies will be summarized in the Safety Analysis Set. The therapies and surgeries with the same sequence/regimen number are counted as one prior therapy/surgery.

Patient data listings of prior anticancer systemic therapies and prior radiotherapies will be provided in the Safety Analysis Set.

## **6.4.5.1 Prior Anticancer Drug Therapies**

The number (percentage) of patients with any prior anticancer therapy, number of prior lines, duration of last prior anticancer systemic therapy, reasons for discontinuation of last anticancer drug therapy, best overall response to the last anticancer drug therapy, time from end of last anticancer drug therapy to first dose date, time from last disease progression to first dose date, and treatment setting will be summarized in the Safety Analysis Set.

## 6.4.5.2 Prior Anticancer Surgeries/ Procedures with Therapeutic Intent

The number (percentage) of patients with any prior anticancer surgery, patients with any prior anticancer procedures, treatment intent of surgeries, treatment intent of procedures, time from last anticancer surgery to first dose, and time from last anticancer procedure to first dose will be summarized in the Safety Analysis Set.

## 6.4.5.3 Prior Radiotherapies

The number (percentage) of patients with any prior radiotherapy, treatment intent, treatment setting, time from end of last radiotherapy to first dose date, and site irradiated will be summarized in the Safety Analysis Set.

#### 6.4.6. Prior and Concomitant Medications

Prior medications are defined as medications that stopped before the first dose of study drugs. Concomitant medications will be defined as medications that 1) started before the first dose of study drugs and were continuing at the time of the first dose of study drugs, or 2) started on or after the date of the first dose of study drugs up to 30 days after the patient's last dose.

Prior and concomitant medications will be coded using the version of World Health Organization Drug Dictionary (WHO DD) drug codes Version B3 March 1, 2022. They will be further classified to the appropriate Anatomical Therapeutic Chemical (ATC) code.

The number (percentage) of patients reporting prior and concomitant medications will be summarized by ATC medication class and WHO DD preferred name in the Safety Analysis Set.

#### 6.4.7. Medical History

Medical History will be coded using Medical Dictionary for Regulatory Activities (MedDRA) Version 25.0. The number (percentage) of patients reporting a history of any medical condition, as recorded on the CRF, will be summarized by System Organ Class and Preferred Term for the Safety Analysis Set.

Patient data listings of medical history will be provided.

# 6.5. Efficacy Analysis

### 6.5.1. Secondary Efficacy Endpoints

The secondary efficacy endpoints (ie, ORR, DCR, PFS, and DOR) assessed by investigators using RECIST v1.1 will be summarized descriptively to evaluate the antitumor activities of sitravatinib in combination with tislelizumab by cohorts.

Efficacy analyses will be provided based on both the Efficacy Evaluable Analysis Set and the Safety Analysis Set. The Efficacy Evaluable Analysis Set will be the primary analysis set for

response analyses; and the Safety Analysis Set will be the primary analysis set for time-to-event analyses. No formal hypothesis testing is planned.

### **ORR** by Investigators

The BOR is the best overall response observed from the date of first dose until disease progression, death, cut-off date, or initiation of post-treatment anticancer therapy, whichever occurs first.

The ORR is defined as the percentage of patients whose BOR is confirmed CR or confirmed PR assessed by investigators per RECIST v1.1. Patients with no post-baseline response assessment (for any reason) will be considered as non-responders. The ORR will be summarized with descriptive statistics and the corresponding two-sided 95% CIs calculated from Clopper-Pearson exact method will be also presented. The primary analysis of ORR is based on Efficacy Evaluable Analysis Set and the sensitivity analysis of ORR is based on the Safety Analysis Set.

ORR based on unconfirmed PR or CR will also be calculated in this study.

## Disease Control Rate and Clinical Benefit Rate by Investigators

DCR is defined as the proportion of patients with BOR as CR, PR, or SD assessed by investigator per RECIST v1.1.

CBR is defined as the proportion of patients with BOR as CR, PR, or SD lasting  $\geq$  24 weeks assessed by investigator per RECIST v1.1.

DCR and CBR assessed by investigators will be analyzed similarly to ORR.

## **Progression Free Survival by Investigators**

PFS is defined as the time from the date of first dose of study drugs to the date of first documentation of disease progression assessed by investigator per RECIST v1.1 or death, whichever occurs first. The primary analysis of PFS is based on Safety Analysis Set and the supplementary analysis of PFS is based on Efficacy Evaluable Analysis Set. The censoring rules for the analysis of PFS are presented in Table 1. Kaplan Meier methodology will be used to estimate median, Q1, and Q3 of PFS, and the event-free rates at 3, 6, 9, and 12 months. 95% CIs for median and other quantiles of PFS will be estimated using the method of Brookmeyer and Crowley (Brookmeyer and Crowley, 1982). And 95% CIs for event-free rates will be estimated using Greenwood's formula (Greenwood, 1926). Kaplan-Meier curves will be constructed to provide a visual description of the PFS change with time.

Table 1: Censoring Rules for Progression-Free Survival Per RECIST Version 1.1

| | Derivation rules | Outcome |
|---|---|---|
| No progression at the time of data cut-off or withdrawal from study or lost to follow up | Date of last adequate radiologic assessment prior to or on date of data cut-off or withdrawal from study or lost to follow up | Censored |
| New anticancer therapy started prior to disease progression or death | Last adequate radiological assessment<br>before the new anticancer therapy<br>(hypothetical strategy) | Censored |

BGB-900-103 09 February 2023 Statistical Analysis Plan 1.0

| No baseline or post-baseline | Date of first dose | Censored |
|---|---|---|
| tumor assessments without death | | |
| within 13 weeks after first dose | | |
| No baseline or post-baseline | Date of death | Event |
| tumor assessments with death | | Event |
| within 13 weeks after first dose | | |
| Death or progression after more | Date of last adequate radiologic | Censored |
| than one missed visit | assessment before missed tumor | Censuled |
| | assessments | |

BeiGene

## **Duration of Response by Investigators**

DOR is defined as the time from the first determination of an objective response until the first documentation of PD as assessed by the investigator per RECIST v1.1, or death, whichever comes first. All the censoring rules for PFS will be applied to DOR. DOR will be analyzed in the responders only. The distribution of DOR, including median, Q1 and Q3, and event-free rates at every 3 months, will be estimated using the Kaplan-Meier method for each treatment group. The 95% CIs for median, Q1, and Q3 of DOR will be estimated using the method of Brookmeyer and Crowley (Brookmeyer and Crowley, 1982). And 95% CIs for event-free rates will be estimated using Greenwood's formula (Greenwood, 1926).

# Time to Response by Investigators

Time to response (TTR) will be summarized using descriptive statistics, such as mean, median, and standard deviation. Only patients who have achieved objective response by investigators per RECIST v1.1 will be included in the analysis of TTR.

#### **Subgroup Analysis**

To determine if the treatment effect is consistent across various subgroups, ORR and DCR by the investigator's review and their 95% CIs will be estimated and plotted within each category of the following subgroups in the efficacy evaluable analysis set.

In cohort A, B, F, H, and I, subgroup variables may include, but not limited to:

- Age ( $< 65 \text{ versus} \ge 65$ )
- Sex (Male versus Female)
- Baseline ECOG (0 versus 1)
- Smoking Status (Current/Former versus Never)
- PD-L1 Tumor Cell Score
  - $\circ$  < 1% versus  $\geq$  1% (cohort A, B, and F)
  - 1%-49% versus  $\geq 50\%$  (cohort H and I)
- Disease Status (Metastatic versus Locally advanced)
- Baseline Tumor Size (At/above median versus Below median)

In cohort E, subgroup variables may include, but not limited to:

BeiGene 09 February 2023

- Age ( $< 65 \text{ versus} \ge 65$ )
- Sex (Male versus Female)
- Baseline ECOG Performance Status (0 versus 1)
- AJCC Disease Stage at Initial Diagnosis
- PD-L1 Tumor Cell Score (< 1% versus  $\ge 1\%$ )

In cohort G, subgroup variables may include, but not limited to:

- Age ( $< 65 \text{ versus} \ge 65$ )
- Sex (Male versus Female)
- Baseline ECOG Performance Status (0 versus 1)
- Histology (Cutaneous, Acral, Mucosal, and Unknown)
- BRAF Mutation Status (Positive, Negative, and Unknown)
- PD-L1 Tumor Cell Score (< 1% versus  $\ge 1\%$ )

For OS and PFS, Kaplan-Meier plot, median survival time and their 95% CI will be provided for the subgroups of tumor cell PD-L1 expression level.

## 6.5.2. Exploratory Efficacy Endpoints

#### **Overall Survival**

OS is defined as the time from first dose date to the documented death date for patients who died prior to or on the clinical cutoff date. For patients who are alive by the clinical cutoff date, OS will be censored at the last known alive date. The last known alive date will be defined as either the clinical data cutoff date for patients who are still on treatment, or last available date showing patients alive or cut-off date whichever comes first for other alive patients.

Every effort should be made to ensure complete death dates. In the rare case, if day of death date is missing, death date is imputed as the max (last available date showing patients alive + 1, first day of month of death date). Death with missing month and/or year will not be imputed for OS analysis. The patient with imputed death date will be considered as an event for OS analysis.

The distribution of OS, including median, Q1, and Q3, and event-free rates at 3, 6, 9, and 12 months, will be estimated using the Kaplan-Meier method for each treatment group. 95% CIs for median, Q1, and Q3 of OS will be estimated using the method of Brookmeyer and Crowley (Brookmeyer and Crowley, 1982). The 95% CIs for event-free rates will be estimated using Greenwood's formula (Greenwood, 1926). Kaplan-Meier survival probabilities over time for each cohort will be plotted.

## **ORR** by investigator per CA-125

CA-125 definitions agreed by GCIG will be referred to calculate the CA-125 response rate. A CA-125 response is defined as at least a 50% reduction in CA-125 levels from a pretreatment sample. The response must be confirmed and maintained by using the next scheduled CA-125 data (at least 28 days). Patients can be evaluated according to CA-125 only if they have a pretreatment sample

that is at least twice the upper limit of the reference range and within 2 weeks before starting the treatment.

The date when the CA-125 level is first reduced by 50% is the date of the CA-125 response. To calculate response, all patients with an initial CA-125 level of at least twice the upper limit of the reference range as eligible and evaluable will be included. In addition, those patients who have a CA-125 response and whose CA-125 level falls to the reference range can be classified as CA-125 complete responder (Table 2).

**Table 2: Measurement of CA-125** 

| CA-125 Level | CA-125 Measurement |
|---|---|
| Baseline CA-125 more than twice upper limit of normal, later reduced by 50% to normal and maintaining for at least 28 days | CR |
| Baseline CA-125 more than twice upper limit of normal, later reduced by 50% but not to normal | PR |
| CA-125 change out of range of PR and PD | Non-PR, non-PD |
| CA-125 increased at baseline returning to normal after treatment, later twice or higher upper limit of normal (2 consecutive measurements at interval of at least 1 week) | PD (date of first evaluation of progression) |
| CA-125 increased at baseline not returning to normal after treatment, later twice or higher the lowest value (2 consecutive measurements at interval of at least 1 week) | PD (date of first evaluation of progression) |
| CA-125 within reference range at baseline, later twice or higher upper limit of normal (2 consecutive measurements at interval of at least 1 week) | PD (date of first evaluation of progression) |

The analysis of CA-125 response rate will be conducted on the CA-125 Evaluable Analysis Set, Efficacy Evaluable Analysis Set, and Safety Analysis Set.

## PFS assessed by investigator per CA -125

PFS per CA-125 is defined as the time from the date of first dose of study drugs to the date of first documentation of PD assessed by the investigator per CA-125 (GCIG working group criteria) or death, whichever occurs first in all patients with ovarian cancer (cohort E). The censor rule of PFS per CA-125 is the same as the censor rule of PFS per RECISIT 1.1. Kaplan-Meier survival probabilities of PFS assessed by investigator per CA-125 over time for each cohort will be plotted.

# 6.6. Safety Analysis

All safety analyses will be performed by cohorts, NSCLC population and total in Safety Analysis Set. Safety and tolerability will be assessed, where applicable, by incidence, severity, and change

from baseline values for all relevant parameters including AEs, laboratory values, vital signs, and ECG findings.

## 6.6.1. Extent of Exposure

The following measures of the extent of exposure will be summarized:

- Duration of exposure (months) for tislelizumab is defined as (last date of exposure first dose date + 1) / 30.4375. For treatment ongoing patients, use cutoff date as the 'last date of exposure'; for patients treated with tislelizumab and discontinued from treatment, 'last date of exposure' is defined as the earliest date of cutoff date, death date and last dose date + 20.
- Duration of exposure (months) for sitravatinib is defined as (last date of exposure first dose date + 1) / 30.4375. For treatment ongoing patients, use cutoff date as the 'last date of exposure'; for patients treated with sitravatinib and discontinued from treatment, use last dose date as 'last date of exposure'.
- Number of treatment cycles received: defined as the total number of treatment cycles in which at least one dose of the study drug is administered.
- Total dose received per patient (mg) is defined as the cumulative dose of the study drug during the treatment period of the study.
- Actual dose intensity (mg/cycle) for tislelizumab is defined as the 21 x total cumulative dose (mg) received by a patient / (last dose date prior to cut off date + 21 first dose date).
- Actual dose intensity (mg/day) for sitravatinib is defined as the cumulative dose (mg) received by a patient divided by duration of exposure (days).
- Relative dose intensity is defined as the actual dose intensity divided by the planned dose intensity x 100. The planned dose intensity is 200 (mg/cycle) for tislelizumab and 120 (mg/day) for sitravatinib.
- Number (%) of patients with dose modifications
- Number (%) of patients with dose reductions and number of dose reductions per patient (sitravatinib only)
- Number (%) of patients with dose interruptions
- Number (%) of patients with dose delay (tislelizumab only)
- Duration of dose interruption (sitravatinib only)

Patient data listings will be provided for all dosing records, and for the above calculated summary statistics.

## 6.6.2. Adverse Events

AEs will be graded by the investigators using NCI-CTCAE Version 5.0. The AE verbatim descriptions (investigator terms from the eCRF) will be classified into standardized medical terminology using MedDRA. AEs will be coded to the MedDRA (Version 25.0 or higher) lowest level term closest to the verbatim term, along with the linked MedDRA Preferred Term (PT) and primary System Organ Class (SOC).

BeiGene 09 February 2023

## **6.6.2.1 Treatment Emergent Adverse Event**

A treatment-emergent adverse event (TEAE) is defined as an AE that had onset or increase in severity level date on or after the date of the first dose of study drug up to 30 days after the last dose (any component of combination treatment whichever is last) or the initiation of subsequent anticancer therapy, whichever comes first. Treatment-related TEAEs include those events considered by the investigator to be related to study drug or with a missing assessment of the causal relationship. Summary tables will generally focus on those TEAEs and treatment-related TEAEs.

The incidence of TEAEs will be reported as the number (percentage) of patients with TEAEs by SOC, PT, and the worst grade. A patient will be counted only once by the highest severity grade within an SOC and PT, even if the patient experienced more than 1 TEAE within a specific SOC and PT. An overall summary and separate summaries of the number (%) of patients with the below types of TEAE will be generated:

#### • All TEAEs

- TEAEs by SOC and PT
- o TEAEs by PT
- Treatment-related TEAEs by SOC and PT
- o Treatment-related TEAEs by PT
- TEAEs related to sitravatinib by SOC and PT
- TEAEs related to tislelizumab by SOC and PT

## Serious TEAEs

- Serious TEAEs by SOC and PT
- Serious TEAEs by PT
- Serious TEAEs related to sitravatinib by SOC and PT
- Serious TEAEs related to tislelizumab by SOC and PT
- o Serious treatment-related TEAEs by SOC and PT

### • TEAEs with NCI-CTCAE grade $\geq$ 3

- TEAEs with grade  $\ge$ 3 by SOC and PT
- TEAEs with grade  $\ge$ 3 by PT
- Treatment-related TEAEs with grade  $\geq$  3 by SOC and PT
- Treatment-related TEAEs with grade  $\geq$  3 by PT
- TEAEs related to sitravatinib with grade  $\geq$  3 by SOC and PT
- TEAEs related to tislelizumab with grade  $\geq$  3 by SOC and PT

#### • TEAEs leading to death

o TEAEs leading to death by SOC and PT

BeiGene 09 February 2023

- o Treatment-related TEAEs leading to death by SOC and PT
- TEAEs leading to treatment discontinuation by SOC and PT
  - o TEAEs leading to treatment discontinuation by SOC and PT
  - o Treatment-related TEAEs leading to treatment discontinuation by SOC and PT
  - o TEAEs leading to treatment discontinuation of sitravatinib by SOC and PT
  - o TEAEs leading to treatment discontinuation of tislelizumab by SOC and PT
- TEAEs leading to treatment modification by SOC and PT
  - TEAEs leading to treatment modification by SOC and PT
  - o TEAEs leading to treatment modification of sitravatinib by SOC and PT
  - o TEAEs leading to treatment modification of tislelizumab by SOC and PT
  - o Treatment-related TEAEs leading to treatment modification by SOC and PT

Patient data listings of all AEs, SAEs, TEAEs leading to death, TEAEs leading to treatment discontinuation or otherwise will be provided.

#### 6.6.2.2 Immune- Mediated Adverse Event

Immune-mediated AEs (imAEs) will be identified from all AEs that had an onset date or a worsening in severity from baseline (pretreatment) on or after the first dose of study drug and up to 90 days from the last dose of tislelizumab, regardless of whether the patient starts a new anticancer therapy. If an imAE occurs outside of the above-mentioned TEAE window, it will not be classified as a TEAE.

An overall summary table and separate summaries of the following incidence of immune-mediated adverse events will be provided:

- imAEs by category and PT
- imAEs by PT
- $imAEs \ge Grade 3$  by category and PT
- Serious imAEs by category and PT
- imAEs leading to treatment discontinuation by category and PT
- imAEs leading to tislelizumab discontinuation by category and PT
- imAEs leading to dose modification by category and PT
- imAEs leading to dose modification of tislelizumab by category and PT
- imAEs leading to death by category and PT

Patient data listings of imAEs will be provided.

#### 6.6.2.3 Infusion-related Adverse Event

All AE terms with the wording "Infusion-Related Reactions" (IRRs) or "Infusion Reaction" will be considered as infusion-related AE. Separate summaries of IRRs and IRRs with NCI-CTCAE grade ≥ 3 will be provided by SOC and PT.

### 6.6.2.4 Death

All deaths and causes of death will be summarized by cohorts, NSCLC population, and total, including those occurred during the study treatment period and those reported during the survival follow-up period after treatment completion/discontinuation.

Patient data listings of deaths will be provided.

## 6.6.3. Laboratory Values

Laboratory safety tests will be evaluated for selected parameters described in Table 3.

Laboratories parameters (e.g., hematology, chemistry, and coagulation) are graded in NCI-CTCAE Version 5.0 will be summarized by shifts from baseline NCI-CTCAE grades to maximum post-baseline grades. In the summary of laboratory abnormalities worsened by  $\geq 2$  Grades (eg, hematology and chemistry), parameters with NCI-CTCAE grading in both high and low directions will be summarized separately. The summary tables will report laboratory assessments up to 30 days of the last dose date. Laboratory parameters for potential Hy's Law for liver injury and abnormal thyroid function will also be summarized.

Patient data listings will be provided as appropriate.

BeiGene 09 February 2023

**Table 3: Clinical Laboratory Assessment** 

| Serum Chemistry | Hematology | Coagulation <sup>a</sup> | Thyroid Function | Urinalysis |
|---|---|---|---|---|
| Alkaline<br>phosphatase | Hematocrit | Prothrombin time or INR | TSH | Glucose |
| Alanine aminotransferase | Hemoglobin | aPTT | Т3 | Protein |
| Aspartate aminotransferase | Platelet counts | | T4 | Blood |
| Albumin | WBC count | | | Ketones |
| Total bilirubin | Lymphocyte count | | | 24-hour protein <sup>d</sup> |
| Direct bilirubin | Neutrophil count | | | |
| Blood urea nitrogen or urea | | | | |
| Potassium | | | | |
| Sodium | | | | |
| Corrected calcium b | | | | |
| Creatinine | | | | |
| Glucose | | | | |
| Lactate dehydrogenase | | | | |
| Total protein | | | | |
| Creatine Kinase (CK) ° | | | | |
| CK-MB ° | | | | |

Abbreviations: aPTT, activated partial thromboplastin time; CK, creatine kinase; CK-MB, creatine kinase cardiac

BeiGene 09 February 2023

isoenzyme; INR, International Normalized Ratio; WBC, white blood cell.

- a. Coagulation tests are required at baseline and subsequently as clinically indicated
- b. If not feasible at the local laboratory, total calcium may be performed instead of corrected calcium.
- c. In the event that CK-MB fractionation is not available, please assess troponin I and/or troponin T instead. If tislelizumab has been permanently discontinued, CK and CK-MB testing is no longer required.
- d. On routine urinalysis, if urine protein is  $\geq 2+$  by dipstick, then obtain a 24-hour urine sample for total protein

## 6.6.4. Vital Signs

The number and percentage of patients satisfying the following conditions of systolic blood pressure at any time post-baseline will be summarized:

- 140 mmHg to 159 mmHg, 160 mmHg to 179 mmHg, or  $\ge$  180 mmHg
- > 0, > 20, > 40, or > 60 mmHg maximum increase from baseline

The number and percentage of patients satisfying the following conditions of diastolic blood pressure at any time post-baseline will be summarized:

- 90 mmHg to 99 mmHg, 100 mmHg to 109 mmHg, or  $\geq$  110 mmHg
- > 0, > 10, > 20, or > 30 mmHg maximum increase from baseline

## 6.6.5. Electrocardiograms (ECG)

The number and percentage of patients satisfying the following QTcF conditions at any time post-baseline will be summarized:

- > 450, > 480, or > 500 msec
- > 30 or > 60 msec maximum increase from baseline

### 6.6.6. Eastern Cooperative Oncology Group (ECOG) Performance Status

A shift table from baseline to worst post-baseline in ECOG Performance Status will be summarized.

# 6.7. Pharmacokinetic Analysis

The PK concentrations will be determined using plasma (sitravatinib) or serum (tislelizumab) samples collected at specified time points within a reasonable variation window.

### 6.7.1. Pharmacokinetic Analysis of Sitravatinib

The first 5 patients per cohort and the 12 patients (6 patients from Australian sites and 6 patients from China sites, regardless of cohort) for SMC safety review will contribute on serial PK samples. All other patients will contribute sparse PK samples.

- Serial PK samples will be collected on timepoints with pre-dose, 0.5 hours, 1 hours, 2 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, and 24 hours on Cycle 1 Day 1 and Cycle 1 Day 21.
- Sparse PK samples will be collected on timepoints with pre-dose and 6 hours on Cycle 1 Day 1, Cycle 2 Day 1, and Cycle 5 Day 1.

Plasma Concentrations will be summarized with descriptive statistics for both serial and sparse PK samples. Concentration versus time will be plotted for patients with serial plasma samples individually and summarized graphically using arithmetic mean plots, respectively in the linear (ie, original) scale and semi-logarithmic scale. PK parameters will be calculated based on the BeiGene Work Instruction. The PK parameters will be summarized with descriptive statistics for the serial PK samples. If data allows, the PK parameters will include:

- AUC<sub>0-t</sub>, area under the plasma concentration-time curve from time zero to the last measurable time point
- AUC <sub>0-tau</sub>, area under the plasma concentration-time curve during the dosing interval.
- AUC<sub>0-inf</sub>, area under the plasma concentration-time curve from time zero to infinity
- C<sub>max</sub>, maximum plasma concentration
- CL/F, clearance after oral administration
- T<sub>max</sub>, time to maximum plasma concentration
- $t_{1/2}$ , terminal elimination half-life
- V<sub>z</sub>/F, the terminal volume of distribution after oral administration
- $R_o$ , observed accumulation ratio determined by the ratios of parameters (AUC<sub>0-tau</sub> and  $C_{max}$ ) at steady state and single dose.

Accumulation ratios for selected PK parameters will be estimated by geometric mean ratios of the parameters at steady state (Cycle 1 Day 21 [C1D21]) and single dose (Cycle 1 Day 1 [C1D1]) in linear mixed effect models. The linear mixed effect model for each selected parameter will include the natural logarithmic-transformed PK parameter as the dependent variable, fixed effect of Day (steady state vs single dose) and random effect of patient as independent variables. Each accumulation ratio will be estimated by applying the exponential function on the difference of least square (LS) means of  $\log(PK_{C1D21})$  and  $\log(PK_{C1D1})$ . Similarly, the 95% CI for an accumulation ratio will be obtained by applying the exponential function on the 95% CI for the mean of  $\log(PK_{C1D21})$  -  $\log(PK_{C1D1})$ . For each of the selected PK parameters, the intra-subject CV will be calculated by  $\sqrt{e^{MSE}-1}$  where MSE is the expected mean square error for within patient variability obtained from the linear mixed effect model. Inter-subject CV will be calculated as  $\sqrt{e^{S^2}-1}$  where  $S^2$  is the estimate of variance for the random effect of patient. For each selected parameter, only patients with valid values at single dose and steady state will be included for analyses of accumulation, intra-subject CV and inter-subject CV.

## 6.7.2. Pharmacokinetic Analysis of Tislelizumab

PK samples for tislelizumab will be collected pre-dose of tislelizumab (-30 min) on Day 1 of Cycles 1, 2, 5, 9 and 17, and post-dose (within 30 min after the end of tislelizumab infusion) on Day 1 of Cycle 1 and Cycle 5, and at EOT visit. Serum Concentrations will be summarized with descriptive statistics.

# 6.8. Immunogenicity Analysis

ADA samples for tislelizumab should be collected Day 1 (Predose of tislelizumab, -30 min) of Cycles 1, 2, 5, 9 and 17, and at the EOT Visit. All samples should be drawn at the same time as the PK blood collection for pre-dose of tislelizumab.

The scope of ADA calculations used for characterizing clinical immunogenicity depend on the incidence and kinetics of detected (ADA). Therefore, not all parameters described below may be derived or additional parameters may be added.

The immunogenicity results will be summarized using descriptive statistics by the number and percentage of subjects who develop detectable ADAs. The incidence of positive and neutralizing ADAs will be reported for ADA-evaluable subjects according to the following definitions:

- ADA-evaluable patient: patients who received at least 1 dose of tislelizumab and for whom both baseline ADA and at least 1 postbaseline ADA results are available.
- Treatment-emergent ADA: The sum of both treatment-boosted and treatment-induced ADA-positive patients. Synonymous with "ADA Incidence".
- Treatment-induced ADA: ADA-evaluable patients that were ADA-negative at baseline and ADA-positive following administration of tislelizumab.
- Treatment-boosted ADA: Baseline-positive ADA-evaluable patient with significant increases (4-fold or higher) in ADA titer after tislelizumab administration.
- Persistent ADA: Treatment-induced ADA detected at two or more sampling time points during the treatment (including follow-up period if any), where the first and last ADA-positive samples (irrespective of any negative samples in between) are separated by a period of 16 weeks or longer; or detected in the last time point.
- Transient ADA: Treatment-induced ADA that is not considered as persistent ADA.
- Neutralizing ADA: patients with positive NAb.

The individual immunogenicity results will also be listed.

Additional ADA analyses (such as the effect of immunogenicity on PK, efficacy, and safety) may be conducted if deemed necessary and will be described in a separate analysis plan.

### 7. INTERIM ANALYSIS

No interim analysis is planned.

#### 8. CHANGES IN THE PLANNED ANALYSIS

Table 4 summarizes the major changes in the planned analyses from the statistical section of the study protocol, including the timing, rational and descriptions of the changes. The changes are all made before database lock and not based on any comparative data.

BeiGene 09 February 2023

**Table 4: Statistical Analysis Plan Changes** 

| SAP<br>version | Approval date | Change made from | Rationale of the change | Description of the change |
|---|---|---|---|---|
| 1.0 | This version | Protocol V3.0 | To clarify the definition of the efficacy evaluable analysis set | 1) Change the "disease progression" from the definition of efficacy evaluable analysis set in the protocol into "clinical disease progression" in the SAP. 2) Change the "death before tumor assessment" from the definition of efficacy evaluable analysis set in the protocol into "early death (within 13 weeks of the first dose date)" in the SAP. |
| 1.0 | This version | Protocol V3.0 | To clarify the pharmacokinetic analysis set of different study drugs | Split the Pharmacokinetic Analysis Set in protocol into Sitravatinib Pharmacokinetic Analysis Set and Tislelizumab Pharmacokinetic Analysis Set in the SAP. |
| 1.0 | This version | Protocol V3.0 | To clarify the specific study drug of the ADA analysis set | Change the name of ADA Analysis Set in protocol into Tislelizumab ADA Analysis Set in the SAP. |
| 1.0 | This version | Protocol V3.0 | For efficacy analysis purpose of the cohort E (OC) | Add the Evaluable for CA-125 Response Set. |
| 1.0 | This version | Protocol V3.0 | For efficacy analysis purpose of the cohort E (OC) | Add an exploratory endpoint: ORR per CA-125. |
| 1.0 | This version | Protocol V3.0 | To align with<br>BeiGene's current<br>standard | The definition of TEAE is different between protocol and SAP. In the protocol, "TEAE classification also applies to irAEs recorded up to 90 days after the last dose of tislelizumab, regardless of whether the patient starts a new anticancer therapy." In this SAP, "If an imAE occurs outside of the above-mentioned TEAE window, it will not be classified as a TEAE". The update of TEAE window streamlines the TEAE derivation so all TEAEs can be identified programmatically instead of relying on the manual medically review of imAE. |
| 1.0 | This version | Protocol V3.0 | To align with<br>BeiGene's current<br>standard | Change the name of immune-related adverse events (irAEs) into immunemediated AEs (imAEs). |

#### 9. REFERENCES

Brookmeyer R, Crowley J. A confidence interval for the median survival time. Biometrics. 1982;38:29-41.

Greenwood M. The Natural Duration of Cancer. Reports on Public health and medical subjects. 1926;33:1-26.

ICH. Addendum on Estimands and Sensitivity Analysis in Clinical Trials to the Guideline on Statistical Principles for Clinical Trials: E9(R1). 2019.

Mantel N, Haenszel W. Statistical Aspects of Analysis of Data from Retrospective Studies of Disease. Journal of the National Cancer Institute. 1959;22:719–748.

Sato T. On the Variance Estimator of the Mantel-Haenszel Risk Difference. Biometrics. 1989; 45:1323–1324.

Common Terminology Criteria for Adverse Events (CTCAE). Version 5.0. United States Department of Health and Human Services, National Institutes of Health, National Cancer Institute, Washington, DC, USA, November 27, 2017.

Eisenhauer EA, T. P. B. J. S. L. S. D. F. R. e. a., 2009. New response evaluation criteria in solid tumours: Revised RECIST guideline (version 1.1). pp. 45:228-47.

Rustin GS, Vergote I, Eisenhauer E, et al., 2011. Definitions for response and progression in ovarian cancer clinical trials incorporating RECIST 1.1 and CA-125 agreed by the Gynecological Cancer Intergroup (GCIG). Int J Gynecol Cancer, pp. 21(2):419-23.

BeiGene Work Instruction. Best Practice Guidance: Non-Compartmental Pharmacokinetic Data Analysis for Clinical Studies. Version 1.0, December 2020.

#### APPENDIX 1. IMPUTATION OF MISSING OR PARTIALLY MISSING DATES

In general, missing or partial dates will not be imputed at the data level. The following rules will apply for the specific analyses and summary purposes mentioned below only.

#### 1.1 Prior/Concomitant Medications/Procedures

When the start date or end date of a medication/therapy/procedure is partially missing, the date will be imputed to determine whether the medication/therapy/procedure is prior or concomitant. The following rules will be applied to impute partial dates for medications.

If start date of a medication/therapy/procedure is partially missing, impute as follows.

- If both month and day are missing, then set to January 01
- If only day is missing, then set to the first of the month
- If the imputed start date > death date, then set to death date

If end date of a medication/therapy/procedure is partially missing, impute as follows.

- If both month and day are missing, then set to December 31
- If only day is missing, then set to last day of the month
- If the imputed end date > death date, then set to death date

If the year of start date or year of end date of a medication/therapy/procedure is missing, or the start date or end date is completely missing, do not impute.

#### 1.2 Adverse Events

The imputation rule for the safety analysis will be used to address the issues with partial dates. When the start date or end date of an adverse event is partially missing, the date will be imputed to determine whether the adverse event is treatment-emergent. When in doubt, the adverse event will be considered treatment-emergent by default. The following rules will be applied to impute partial dates for adverse events:

If year of the start date is missing or start date is completely missing, do not impute. Impute AE end date first if both AE start date and end date are partially missing. If year of the end date is missing or end date is completely missing, do not impute.

If end date of an adverse event is partially missing, impute as follows.

- If both month and day are missing, then set to December 31
- If only day is missing, then set to last day of the month
- If the imputed end date > death date, then set to death date

If start date of an adverse event is partially missing, impute as follows.

- If both month and day are missing and year = year of treatment start date, then set to treatment start date
- If both month and day are missing and year  $\neq$  year of treatment start date, then set to January

01

- If day is missing and month and year = month and year of treatment start date, the set to treatment start date
- If day is missing and month and year ≠ month and year of treatment start date, the set to first of the month
- If the imputed AE start date is after AE end date (maybe imputed), then update AE start date with AE end date as final imputed AE start date
- If the imputed start date > death date, then set to death date

### 1.3 Disease history and prior therapy (Drug, surgery/procedure, radiotherapy)

For prior therapy, impute end date first.

If end date of a prior therapy is partially missing, impute as follows.

- If both month and day are missing, then set to December 31
- If only day is missing, then set to last day of the month
- If the imputed end date > first dose date, then set to first dose date -1

If start date of a prior therapy is partially missing, impute as follows.

- If both month and day are missing, then set to January 01
- If only day is missing, then set to the first of the month
- If the imputed start date > end date, then set to end date

The following rules will be applied to impute partial dates such as initial diagnosis date, initial BCLC staging date, relapse date, therapy date (start/end date), or surgery date etc.

If date of a disease history is partially missing, impute as follows.

- If both month and day are missing, then set to January 01
- If only day is missing, then set to the first of the month
- If the imputed date > first dose date, then set to first dose date -1

If diagnosis date of metastatic disease/locally advanced is partially missing, impute as follows.

- If both month and day are missing, then set to January 01
- If only day is missing, then set to the first of the month
- If the imputed date > first dose date, then set to first dose date -1
- If the imputed date < (imputed) date of initial diagnosis date, then set to initial diagnosis date.

If the date of response to prior therapy is partially missing, impute as follows.

- If both month and day are missing, then set to January 01
- If only day is missing, then set to the first of the month

BeiGene 09 February 2023

- If the imputed date > first dose date, then set to first dose date -1
- If the imputed date < the start date of prior therapy, then set to the start date of prior therapy +1.

## 1.4 Subsequent anti-cancer therapy

If start date of subsequent anti-cancer therapy is partially missing, impute as follows.

- If both month and day are missing, then set to December 31
- If only day is missing, then set to last day of the month
- If the imputed start date > min (death date, data cutoff date, study discontinuation date, start date of the next subsequent therapy), then set it as min (death date, data cutoff date, study discontinuation date, start date of the next subsequent therapy)

If stop date of is partially missing, impute as follows.

- If both month and day are missing, then set to December 31
- If only day is missing, then set to last day of the month
- If the imputed stop date > min (death date, data cutoff date, study discontinuation date, start date of the next subsequent therapy), then set it as min (death date, data cutoff date, study discontinuation date, start date of the next subsequent therapy)
- The (imputed) stop date must be after or equal to the (imputed) start date

If year of the start date/stop date is missing, do not impute.

BeiGene 09 February 2023

#### APPENDIX 2. RULES FOR IDENTIFYING MISSING TUMOR ASSESSMENTS

Identifying two missing tumor assessments

- 1) Input scheduled TA visit list
  - a. (6wk-12wk-18wk-24wk-30wk-36wk-42wk-48wk) for this study with TA as every 6 weeks for the first 12 months (52 weeks), then every 9 weeks thereafter
- 2) Identify last evaluable TA before PD or death (LPTADT) and map it to the closest scheduled visit (LPTADT WK).
  - a. In the event of unscheduled TA, choose the closest scheduled visit number (e.g. 6wk) as LPTADT\_WK. It can be achieved programmatically by following the classification rule (e.g. defining thresholds) depicted in Table 5 below. (The team can consider mapping all tumor visits if the scheduled visits are uncleaned or questionable)
  - b. Otherwise, assign the scheduled visit number (assuming it is coded correctly) to LPTADT WK
- 3) Find the 2nd TA visit after LPTADT\_WK according to the list in step 1 (LPTADT\_WK\_2)
  - a. If LPTADT\_WK\_2+1wk (assuming 1 week TA window) < earliest of PD/death date, then censor PFS at the LPTADT
  - b. Otherwise, PFS event at the earliest of PD/death date

Table 5 shows how to assign unscheduled TA to a schedule visit. The threshold column is defined as the mid-point between current and next visit (except for baseline); it is the upper limit for LPTADT to be mapped to the prior scheduled assessment (step 2a above). For example, if LPTADT is Week 44 for an unscheduled visit, it will be mapped to Week 42 TA since it is within the threshold for Week 42. Assuming it is SD and the subsequent TA of the patient is PD after Week 58, PFS will be censored at LPTADT (Week 44); had the PD occurred prior to Week 58, it would be counted as an PFS event.

Table 5: Example of Scheduled Tumor Assessments With Time Window

| Weeks | Scheduled week -1 | Scheduled week | Scheduled week+1 | Threshold |
|---|---|---|---|---|
| Baseline | | Baseline | | |
| Every 6 weeks<br>for the first 52<br>weeks | Week 5 | Week6 | Week 7 | Week 9 |
| | Week 11 | Week 12 | Week 13 | Week 15 |
| | Week 17 | Week 18 | Week 19 | Week 21 |
| | Week 23 | Week 24 | Week 25 | Week 27 |
| | Week 29 | Week 30 | Week 31 | Week 33 |
| | Week 35 | Week 36 | Week 37 | Week 39 |
| | Week 41 | Week 42 | Week 43 | Week 45 |
| | Week 47 | Week 48 | Week 49 | Week 52 |
| Every 9 weeks thereafter | Week 56 | Week 57 | Week 58 | Week 61 |
| | Week 65 | Week 66 | Week 67 | Week 70 |
| | Week 74 | Week 75 | Week 76 | |